CLINICAL TRIAL: NCT07243080
Title: Comparison Between the Efficacy of Rivaroxaban vs Enoxaparin in Post-Operative Deep Venous Thrombosis Prophylaxis After Exploratory Laparotomy
Brief Title: Comparative Efficacy of Rivaroxaban and Enoxaparin in Post-Laparotomy DVT Prevention
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Hospital Lahore (Other)
Collaborators: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Mashhood Ahmad Shad, Principle Investigator, Mayo Hospital Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DRSHAD-GS-2025-001
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Deep Venous Thromboses; Laparotomy Patients
Keywords: Deep Vein Thrombosis; Exploratory Laparotomy; Rivaroxaban; Enoxaparin; Venous Thromboembolism; Anticoagulation; Prophylaxis; Randomized Controlled Trial; Thromboprophylaxis
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Intervention Model Description: This randomized, parallel-group, Phase 4 clinical trial enrolled a total of 212 adult patients undergoing emergency exploratory laparotomy at Mayo Hospital, Lahore. Participants were allocated in a 1:1 ratio to one of two arms:
  Arm 1: Rivaroxaban 10 mg orally once daily for 7 days
  Arm 2: Enoxaparin 40 mg subcutaneously once daily for 7 days
  Allocation was performed using a computer-generated randomization sequence with concealment via sealed opaque envelopes. The trial used single masking (outcomes assessor blinded); the radiologist performing duplex ultrasonography and the data analyst were blinded to group allocation.
  The study compared the two interventions in parallel to evaluate the incidence of postoperative deep vein thrombosis (DVT) on days 5 and 10, as detected by duplex color Doppler ultrasound.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rivaroxaban Group (Active Comparator): Arm 1 Title: Rivaroxaban Group Arm Type: Experimental Intervention Name: Drug: Rivaroxaban Descri
  Interventions: Drug: rivaroxaban (10mg)
- Enoxaparin Group (Active Comparator): Arm 2 Title: Enoxaparin Group
  Arm Type: Active Comparator
  Intervention Name: Drug: Enoxaparin
  Description: Participants receive enoxaparin 40 mg subcutaneously once daily for 7 days after emergency exploratory laparotomy, in addition to standard perioperative care and mechanical prophylaxis.
  Interventions: Drug: Enoxaparin 40 mg SC

INTERVENTIONS:
Drug: rivaroxaban (10mg) — Name: Drug: Rivaroxaban
  Type: Drug
  Description: Participants receive rivaroxaban 10 mg orally once daily for 7 days following emergency exploratory laparotomy. All patients also receive standard perioperative management and mechanical prophylaxis as per institutional guidelines.
  Other Names: Xarelto
  Arms: Rivaroxaban Group
Drug: Enoxaparin 40 mg SC — Name: Drug: Enoxaparin
  Type: Drug
  Description: Participants receive enoxaparin 40 mg subcutaneously once daily for 7 days following emergency exploratory laparotomy. All patients also receive standard perioperative management and mechanical prophylaxis as per institutional guidelines.
  Other Names: clexane
  Arms: Enoxaparin Group

SUMMARY:
The goal of this clinical trial is to learn if rivaroxaban works better than enoxaparin to prevent deep vein thrombosis (DVT) after emergency exploratory laparotomy in adults. It will also learn about the safety of rivaroxaban compared to enoxaparin.

The main questions it aims to answer are:

Does rivaroxaban lower the number of patients who develop DVT after exploratory laparotomy compared to enoxaparin?

What medical problems or side effects do participants have when taking rivaroxaban versus enoxaparin?

Researchers will compare rivaroxaban (an oral anticoagulant) to enoxaparin (a subcutaneous injection) to see which drug works better to prevent blood clots after surgery.

Participants will:

Take rivaroxaban 10 mg orally once daily for 7 days, or enoxaparin 40 mg subcutaneously once daily for 7 days after surgery

Undergo duplex color Doppler ultrasound scans of the legs on day 5 and day 10 after surgery

Be monitored for bleeding, complications, and other side effects

DETAILED DESCRIPTION:
Postoperative venous thromboembolism (VTE), which includes deep vein thrombosis (DVT) and pulmonary embolism (PE), is a major and preventable cause of morbidity and mortality after surgery. Patients undergoing emergency exploratory laparotomy are at especially high risk due to prolonged operative times, systemic inflammation, and immobility. While low-molecular-weight heparins (LMWH), such as enoxaparin, are the current standard for prophylaxis, direct oral anticoagulants such as rivaroxaban offer potential advantages in terms of ease of administration, compliance, and patient comfort.

This randomized controlled trial was designed to compare the efficacy and safety of once-daily oral rivaroxaban (10 mg) with once-daily subcutaneous enoxaparin (40 mg) in preventing postoperative DVT in adult patients undergoing emergency exploratory laparotomy at Mayo Hospital, Lahore.

Eligible patients were adults aged 18-80 years undergoing emergency laparotomy for traumatic or non-traumatic indications and expected to remain immobile for more than 24 hours postoperatively. Patients with pre-existing DVT, morbid obesity (BMI ≥40), active bleeding risk, mechanical ventilation, myocardial infarction, cerebrovascular accident, or current anticoagulation therapy were excluded.

Participants were randomized using a computer-generated sequence with allocation concealment. Rivaroxaban or enoxaparin was given for 7 days postoperatively, in addition to standard perioperative care and mechanical prophylaxis.

The primary outcome was the incidence of DVT as confirmed by duplex color Doppler ultrasound on postoperative days 5 and 10. Any noncompressible or indistinct venous segment was scored as positive for DVT. Wells scores were also recorded to stratify risk.

The secondary outcomes included bleeding complications, duration of hospital stay, time to ambulation, and cost comparison between the two regimens. Safety assessments focused on clinically significant bleeding events and other adverse reactions.

A total of 212 patients were enrolled (106 in each arm). On day 5, rivaroxaban showed a significantly lower rate of DVT compared to enoxaparin (3.8% vs 12.3%). By day 10, the difference remained significant (8.5% vs 20.8%). Wells scores showed no significant differences between groups. No major bleeding events were reported in either arm.

The findings suggest that rivaroxaban is more effective than enoxaparin in reducing postoperative DVT after emergency exploratory laparotomy without increasing bleeding risk. These results add evidence that rivaroxaban may be a safe and convenient alternative to LMWH for high-risk general surgical patients. However, larger multicenter trials with longer follow-up are needed to confirm safety and evaluate long-term outcomes such as pulmonary embolism and late-onset DVT.

ELIGIBILITY:
Inclusion Criteria:• Patients aged 18 to 80 years

* Both male or female patients
* Patients who have undergone emergent exploratory laparotomy for any reason whether traumatic or non-traumatic
* Patients with expected immobility for more than 24 hours

Exclusion Criteria:

* Patients with diagnosed pre-operative DVT
* BMI more than 40
* Patient who are on mechanical ventilation post operatively
* Patient with postoperative Myocardial infarction, ischemic heart disease or cerebrovascular accident
* Patients who have undergone limb surgery in addition to exploratory laparotomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Deep Vein Thrombosis (DVT) | Postoperative Day 5 and Day 10
  Presence of DVT in the lower limbs will be assessed by duplex color Doppler ultrasonography on postoperative day 5 and day 10. A noncompressible or indistinct venous segment on ultrasound will be considered positive for DVT. The outcome will be reported as the proportion of participants in each treatment arm who develop DVT.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Uzair Qureshi, FCPS, Study Chair — Mayo Hospital Lahore
Locations (1):
- Mayo Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected during the trial (including demographics, clinical variables, Wells scores, ultrasound results, and outcomes) will not be made publicly available. Only aggregated results will be reported in publications and presentations.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT07243080/Prot_SAP_ICF_000.pdf